CLINICAL TRIAL: NCT05174299
Title: The Effect of Multi-target Magnetic Stimulation on Freezing Gait in Parkinson's Disease
Brief Title: The Effect of Multi-target Magnetic Stimulation on Freezing Gait in PD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Kezhong Zhang, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-SR-209
Record Dates: First submitted 2021-11-08; First posted 2021-12-30 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: freezing of gait; Therapeutics; rTMS; spinal cord stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- double active magnetic stimulation (Experimental): the multi-target magnetic stimulation on motor cortex combined with spinal cord
  Interventions: Device: magnetic stimulation
- single active magnetic stimulation (Active Comparator): the active magnetic stimulation on motor cortex and sham stimulation on spinal cord
  Interventions: Device: magnetic stimulation
- double sham magnetic stimulation (Sham Comparator): the sham magnetic stimulation on motor cortex and sham stimulation on spinal cord
  Interventions: Device: magnetic stimulation

INTERVENTIONS:
Device: magnetic stimulation — For Experimental Arm, active magnetic stimulation on motor cortex followed by active magnetic stimulation on spinal cord, patients underwent ten sessions of double active magnetic stimulation with low frequency repetitive transcranial magnetic stimulation (rTMS) over the bilateral primary motor cortex of the lower leg followed by low frequency repetitive magnetic stimulation over the spinal cord. For Active Comparator Arm, active magnetic stimulation on motor cortex followed by sham magnetic stimulation on spinal cord. For Sham Comparator Arm, sham magnetic stimulation on motor cortex followed by sham magnetic stimulation on spinal cord.

SUMMARY:
This study is a double-blinded randomized study examining the effectiveness of the multi-target magnetic stimulation treatment on Freezing of Gait (FOG) phenomenon in patients with Parkinson's disease. We hypothesize that treatment using magnetic stimulation on motor cortex combined with spinal cord will improve FOG and gait symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Patients in the Experimental group underwent ten sessions of double active magnetic stimulation with low frequency repetitive transcranial magnetic stimulation (rTMS) over the bilateral primary motor cortex of the lower leg followed by low frequency repetitive magnetic stimulation over the spinal cord, whereas patients in the Active Comparator group underwent ten sessions of single active magnetic stimulation with low frequency rTMS over the bilateral primary motor cortex of the lower leg. In addition, patients in the Sham Comparator group underwent 10 sessions of double sham rTMS on motor cortex and spinal cord. Assessments of FOG, gait function, motor symptoms and excitability of primary motor cortex motor were performed three times: at baseline, one day post intervention, one month post intervention.

ELIGIBILITY:
Inclusion Criteria:

* 1.Idiopathic Parkinson's disease (PD), as diagnosed by a neurologist.
* 2.Item 3 of the Freezing of Gait Questionnaire(FOG-Q) scored ≥1.
* 3.Age between 40 and 80 years old.
* 4.Mini-Mental State Examination score >24.
* 5.Ability to walk 30 meters independently.
* 6.Stable medication.
* 7.Patients experienced FOG in both medication "on" and "off" states.

Exclusion Criteria:

* 1.Other neurological or psychiatric disorders.
* 2.Severe personality disorder.History of epilepsy, seizures, or convulsions.
* 3.History of head injury or stroke.
* 4.Metal remains of the skull or inside the brain (outside the oral cavity).
* 5.Surgeries including metallic implants or known history of metal particles in the eye, pacemakers,hearing devices transplantation, or medical pumps.
* 6.Severe dyskinesia, termor, cognitive, visual or auditory impairment.
* 7.Patients who could not complete the follow-up.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes of Freezing of Gait Questionnaire (FOG-Q) | Assessed at baseline, one day post intervention, one month post intervention
  The Freezing of Gait questionnaire will be used to quantify the frequency and severity of this symptom. The score will be compared to the baseline. The minimum and maximum values of the FOG-Q are 0 and 24. A higher FOG-Q score means a worse outcome.

SECONDARY OUTCOMES:
The motor part of the Unified Parkinson's Disease Rating Scale | Assessed at baseline, one day post intervention, one month post intervention
  The measure mainly reflects the overall severity of Parkinson's disease motor symptoms. The minimum and maximum values of the motor part of the Unified Parkinson's Disease Rating Scale are 0 and 108. A higher score means a worse outcome.
Gait speed | Assessed at baseline, one day post intervention, one month post intervention
  Gait speed (m/s) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test.
Stride length | Assessed at baseline, one day post intervention, one month post intervention
  Stride length (cm) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test.
Stride time variability | Assessed at baseline, one day post intervention, one month post intervention
  Stride time variability (%) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test.
  Stride time variability was expressed as coefficient of variation [CV].
Double support | Assessed at baseline, one day post intervention, one month post intervention
  Double support (%) was evaluated at baseline, one day post intervention, one month post intervention using a portable Inertial Measurement Unit system during a 5-m timed Up-and-Go (TUG) test.
Resting motor threshold (RMT) | Assessed at baseline, one day post intervention.
  RMT (% TMS output intensity) is defined as the lowest intensity required to elicit MEPs of > 50 μV in at least 5 of 10 consecutive trials while the target muscle is relaxed. RMT was determined to be the nearest 1% of the maximum stimulator output.
MEP amplitude at 120% RMT intensity (AMP) | Assessed at baseline, one day post intervention.
  Five single stimuli were delivered to the optimal stimulation point at an intensity of 120% of RMT, and the mean peak-to-peak amplitude of the MEPs was calculated, which is the AMP (mV).
Cortical silent period (CSP) | Assessed at baseline, one day post intervention.
  The CSP (ms) is measured through electromyographic signal recording (EMG) on a target muscle and refers to the period of EMG silence following the elicitation of a motor-evoked potential (MEP) through a single TMS pulse delivered over the contralateral primary motor cortex.
  Individuals were asked to actively contract abductor pollicis brevis (APB) with 20% of the maximum force, while a single pulse with 150% of RMT was applied to the opposite primary motor cortex. We recorded the time from pulse outputting to the recovery of inhibited active contraction as CSP. The above protocol was repeated ten times, and the average value of CSP was calculated.
Short-interval intracortical inhibition (SICI) | Assessed at baseline, one day post intervention.
  SICI was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with a 4ms interstimulus interval between conditioning and test stimuli. Ten trials were acquired for each interstimulus interval. SICI was expressed as the percentage ratio between the test and conditioning MEP.
Intracortical facilitation (ICF) | Assessed at baseline, one day post intervention.
  ICF was assessed with a subthreshold conditioning stimulus (80% RMT) and a supra-threshold test stimulus (1 mV MEP) with a 15 ms interstimulus interval between conditioning and test stimuli. Ten trials were acquired for each interstimulus interval. ICF was expressed as the percentage ratio between the test and conditioning MEP.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No